CLINICAL TRIAL: NCT05956704
Title: The Effectiveness and Safety of Different Design of Orthokeratology Lenses to Reduce Myopia Growth
Brief Title: The Different Design of Orthokeratology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2023031
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental)
  Interventions: Device: Orthokeratology with aspheric wide inversion zone design in the optical zone
- Control group (Active Comparator)
  Interventions: Device: Orthokeratology with traditional spherical design in the optical zone
- Blank control group (No Intervention)

INTERVENTIONS:
Device: Orthokeratology with aspheric wide inversion zone design in the optical zone — An orthokeratology lens with an altered optical zone design is designed for an aspherical wide inversion arc in the optical zone
  Arms: Experimental Group
Device: Orthokeratology with traditional spherical design in the optical zone — Subjects wore the orthokeratology with traditional spherical design in the optical zone
  Arms: Control group

SUMMARY:
In this study, we intend to enroll orthokeratology subjects aged 8-18 years old with binocular myopia up to and including -4.00 D. They were randomly selected to wear both orthokeratology of different designs, one with an aspheric wide inversion zone design in the optical zone and the other with a traditional spherical curved segment design, and to investigate the differences between these two lenses in terms of their effectiveness in myopia retardation, defocus, and aberration.

ELIGIBILITY:
Inclusion Criteria:

* The age is greater than 8 years and less than 18 years
* The myopia was within -4.00D (including -4.00D), and the astigmatism was within 1.50D (including 1.50D) in both eyes.
* Be able to complete 12 months of follow-up
* They were able to understand the purpose of the trial, volunteered to participate, and signed informed consent by the subjects themselves or their legal guardians

Exclusion Criteria:

* One eye met the inclusion criteria
* Patients with systemic diseases causing immunocompromised or affecting orthokeratology
* There are other eye diseases that affect orthokeratology lens wearing, such as dacryocystitis, blepharitis, various inflammation, glaucoma, etc
* Abnormal cornea
* Previous corneal surgery or corneal trauma history
* Active keratitis (e.g., corneal infection)
* Patients with best corrected distance visual acuity of less than 5.0
* Patients with corneal flat curvature lower than 39.00D, or higher than 48.00D
* Patients with refractive instability
* Patients with overt strabismus
* The corneal epithelium showed obvious fluorescent staining, which was not suitable for patients wearing orthokeratology lenses
* Patients with dry eye are not suitable for orthokeratology
* Patients with corneal endothelial cell density less than 2000 cells /mm2
* Patients who had worn rigid contact lenses (including orthokeratology lenses) within the previous 30 days

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in axial length | The change of baseline and 1years
  Axial length was measured with a biometer

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No